# Unveiling Follicular Lymphoma Clinical Trials: Analyzing Patient Engagement Patterns and Participation Trends

Obtaining Informed Consent from Follicular Lymphoma Patients: A Document for <a href="Power Clinical Trial's">Power Clinical Trial's</a> Observational Study

Date: September 15, 2023

The Importance of This Informed Consent Form

When you are requested to complete this form, it suggests that you may be eligible to participate in a customized observational clinical research created exclusively for people with follicular lymphoma. This paper serves as a complete guide, revealing the study's key objectives, complex execution strategy, and numerous outcomes, both good and potentially negative. Prior to making a decision, it is critical to properly investigate the intricacies of your possible participation, and receiving advice from a reliable source can give crucial insights. If any aspect of this text is unclear or if you have any queries, please be aware that the researcher is accessible to provide answers.

The Importance of Follicular Lymphoma-Focused Clinical Research

Follicular lymphoma (FL) is a type of non-Hodgkin lymphoma (NHL), which is a cancer that originates in the lymphatic system, a part of the body's immune system. Follicular lymphoma is characterized by the abnormal growth of B-lymphocytes, a type of white blood cell, and typically arises in the lymph nodes, although it can also affect other lymphoid tissues. It is one of the indolent (slow-growing) subtypes of non-Hodgkin lymphoma.

Clinical trials that specifically target follicular lymphoma are essential in assessing the safety and efficacy of emerging treatments for this condition. These trials serve as a critical yardstick for determining whether new drugs outshine traditional therapies, offering robust substantiation for their widespread adoption.

What sets this study apart is its unique focus on the perspectives of individuals coping with follicular lymphoma as they actively participate in a clinical trial incorporating medicinal treatments. The primary emphasis lies in a thorough examination of trial completion rates and voluntary withdrawals within this specific patient cohort.

#### Exploring the Significance of Observational Studies

By participating in this medical trial, you will immerse yourself in an observational study—a unique facet of clinical research designed meticulously to gather insights through unaltered observations of patients while preserving their treatment plans. Researchers will solely observe your journey, methodically assessing the outcomes of your condition without any interventions. This specific trial design plays a crucial role in enhancing our comprehension of the natural progression of a particular medical ailment and its implications for individuals affected by it. Your active participation in this observational study transforms you into a significant contributor, expanding the horizons of medical knowledge and propelling advancements in the care provided to those grappling with the same condition.

## Distinguishing This Trial Among Follicular Lymphoma Clinical Trials

Grasping the uniqueness of this research endeavor holds paramount importance. It operates solely on an observational basis, implying that your participation will not entail any specific treatments or interventions. To make an informed decision regarding potential involvement in a clinical trial, it is crucial to understand the spectrum of follicular lymphoma clinical trials, encompassing interventional studies where participants follow distinct treatment protocols.

Making a well-informed choice about your potential participation in a clinical trial requires an active approach that involves research and comparison of various trials. Resources like Clinicaltrials.gov and similar platforms offer a wealth of information on research related to follicular lymphoma. Additionally, Power's dedicated web platform presents a comprehensive list of ongoing follicular lymphoma clinical trials actively seeking volunteers. Equipping yourself with thorough research and a comprehensive

understanding of different clinical trial types empowers you to confidently shape your participation decision.

#### Active Participation in Clinical Trial Surveying

We extend a heartfelt invitation for you to actively contribute your insights within the context of this observational clinical investigation. This undertaking involves the periodic completion of questionnaires every two weeks, requiring approximately 20-30 minutes of your valuable time. Additionally, we are fully prepared to conduct check-in calls at quarterly intervals, a practice that will be upheld throughout your participation in the trial.

It is imperative to underscore that your engagement in the trial's survey phase is entirely at your discretion. You have the liberty to decide whether to respond to specific questions or complete the entire questionnaire. Moreover, you have the prerogative to discontinue your participation in the trial at any point, should you deem it necessary. Recognizing that the decision to enroll in a clinical study is deeply personal, we are dedicated to offering the appropriate support. Your privacy and comfort are fundamental to us, and we are unwavering in our commitment to respecting and facilitating your decision-making process throughout the trial.

### Safeguarding the Privacy of Your Responses

Ensuring the absolute privacy of your information remains a top priority throughout the entire duration of this clinical trial. To protect your anonymity, we kindly urge you to refrain from disclosing any personal or identifiable details in your questionnaire responses. The dedicated research team is unwavering in their commitment to enhancing the security of your privacy. However, it's important to acknowledge that certain legal circumstances may arise, requiring the disclosure of your data.

# Acknowledging Potential Health Concerns

Despite the notable progress achieved through clinical trials, it remains imperative to recognize the potential health concerns that participants may confront, particularly in investigations of novel medications.

Nevertheless, our observational clinical research adopts a distinct approach, deliberately minimizing these concerns by refraining from the use of experimental therapies in individuals. Our principal objective is centered on meticulous monitoring and comprehensive outcome evaluation, with the utmost commitment to averting any unnecessary health risks.

#### Potential Advantages

While participants in this observational clinical research may not experience immediate benefits, their involvement holds the potential to impact others significantly. The data gathered from participants will contribute to enhancing future approaches to enrolling individuals with follicular lymphoma, potentially expanding the realm of medical research. Those who embark on this therapeutic journey have the capacity to ignite substantial change within the field of medical research, potentially shaping the course of follicular lymphoma patients.

Setting Sail on the Quest for Inclusivity in Clinical Trials

A plethora of online resources stand ready for your active engagement if you are fueled by an insatiable curiosity to explore the nuanced landscape of diversity in clinical trials.

Whether you aim to comprehend the complexities of the barriers and potentialities associated with diversity in clinical research or to broaden your perspectives, the following resources could serve as invaluable guides:

Gross, Annette S., Anya C. Harry, Christine S. Clifton, and Oscar Della Pasqua.

"Clinical trial diversity: An opportunity for improved insight into the determinants of variability in drug response." *British Journal of Clinical Pharmacology* 88, no. 6 (2022): 2700-2717.

Charrow, Alexandra, Fan Di Xia, Cara Joyce, and Arash Mostaghimi. "Diversity in dermatology clinical trials: a systematic review." *JAMA dermatology* 153, no. 2 (2017): 193-198.

Affirmation of Informed Participation

I affirmatively acknowledge that I have invested ample time in comprehending and internalizing the information contained in the informed consent form. This understanding has been attained through either independent examination or with the guidance of a trusted individual who has conveyed its essence to me. All of my inquiries and apprehensions have been addressed comprehensively to my full satisfaction.

I am fully aware that my involvement in this study is a product of my personal choice, and I maintain the exclusive right to revoke my consent without the necessity of providing justification or incurring financial obligations. It has been made clear to me that a copy of this informed consent form will be provided for my personal records.

Following thorough consideration and a comprehensive review of all the materials furnished to me, I hereby grant my approval to participate in this study, affirming my informed and self-governing decision.

| Participant Name |
|-----------------------|
| Participant Signature |
| Date |

Confirmation by an Informed Consent Facilitator

I certify that I had a full conversation with the participant, meticulously clarifying the complexities included within this written content. My goal was to ensure that the participant had a thorough awareness of the research's principal objectives, methods, potential risks and benefits, and other essential components of the follicular lymphoma clinical study.

The participant was given considerable time for inquiry, which facilitated the creation of questions and the explanation of concerns or misconceptions. It is critical to emphasize

| that participation in this study is fully | voluntary, and participants have the unlimited right |
|---|---|
| to leave at any time, for any reason, | without incurring any financial responsibilities. |

Following the granting of consent by the participant, a meticulously preserved replica of this written document was provided to them, functioning as a repository for their personal information.

| Printed Name of Assisting Researcher |
|--------------------------------------|
| Signature of Assisting Researcher |
| Date |